CLINICAL TRIAL: NCT00704639
Title: A Phase II Study of Cetuximab, Carboplatin and Radiotherapy for Locally Advanced Head and Neck Squamous Cell Carcinoma
Brief Title: Chemoradiation Treatment for Head and Neck Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Trans Tasman Radiation Oncology Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TROG 07.04
Record Dates: First submitted 2008-06-22; First posted 2008-06-25 (Estimated); Last update posted 2017-07-12 (Actual); Status verified 2017-07

CONDITIONS: Head and Neck Cancer
Keywords: Head and Neck; Cetuximab; Carboplatin; Radiotherapy
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Cetuximab; Carboplatin; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single arm (Experimental): Chemoradiation (Cetuximab, Carboplatin and Radiotherapy)
  Interventions: Drug: Cetuximab; Drug: Carboplatin; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Cetuximab — Patients will receive weekly intravenous cetuximab (initial dose 400mg/m2 in the week prior to commencing radiotherapy, then weekly 250mg/m2)for the duration of the radiotherapy
  Other Names: Erbitux
Drug: Carboplatin — Weekly intravenous carboplatin (AUC 2) for the duration of the RT
  Other Names: Paraplatin
Radiation: Radiotherapy — The radiotherapy schedule will be the "infield boost" (IFB) regimen, that is 66 Gy in 35 fractions over 5 weeks: daily for 3 weeks, then twice daily for 2 weeks (or 70 Gy in 35 fractions over 7 weeks for a specific subgroup of patients where IFB is not recommended).

SUMMARY:
This is a Phase II study of cetuximab, carboplatin and radiotherapy (RT) in patients with Locally Advanced Head and Neck Carcinomas (LAHNC) who are unfit for cisplatin.

The aim of this study is to show the feasibility and safety profile of the combination of cetuximab, carboplatin and RT in treatment of patients with LAHNC.

DETAILED DESCRIPTION:
Secondary objectives are to estimate failure free survival (FFS) and overall survival, to evaluate the time to local and regional failure and to determine the site of first failure (characterised as local, regional, distant or combinations). Acute and late treatment toxicities will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated SCC of the oropharynx, larynx or hypopharynx.
* Stage III or IV, excluding T1N1, and metastatic disease (to be confirmed by a chest CT, and abdominal CT or ultrasound scan if patients with abnormal liver function tests or a bone scan or FDG-PET if patients with bone pain).
* Histologically or cytologically confirmed HNSCC
* Disease must be considered potentially curable by chemoradiation
* Patients medically unfit for cisplatin chemotherapy due to one or more of the following reasons:

  * Clinically significant sensori-neural hearing impairment (audiometric abnormalities without corresponding clinical deafness will not be regarded as a contraindication to cisplatin)
  * Severe tinnitus
  * Renal impairment (GFR < 60ml/min)
  * Peripheral neuropathy > grade 2
  * Inability to tolerate intravenous hydration eg due to cardiac disease
  * Co-morbidities (based on clinical judgement by the investigator) associated with ECOG PS 2 that in the view of the investigator would preclude the safe administration of cisplatin
* Performance status ECOG 0, 1 or 2.
* Adequate haematological, renal and hepatic functions as defined by:

  * Absolute neutrophil count (ANC, segmented cells (segs) + bands)>= 1.5 x 109/L
  * Platelet count >= 100 x 109/L
  * Total bilirubin <= 1.5 x upper normal limit
  * Alanine aminotransferase <= 2.5 x upper normal limit
  * Calculated creatinine clearance > 40ml/min (Cockcroft-Gault formula).
  * If calculated creatinine clearance < 50 ml/min, glomerular filtration rate to be measured with DTPA or EDTA scan. If < 40 ml/min not eligible.
* Age >18 years
* Signed written consent
* Suitable for follow-up for 4 years in the view of the investigator

Exclusion Criteria:

* Distant metastases, i.e., any metastatic disease below the clavicles. Patients with lung nodules >10mm will be excluded unless non-malignancy aetiology is established. Patients with lesions 5-10mm can be included if a FDG-PET scan is negative and the investigator considers on clinical grounds that metastasis is unlikely. Patients with lesions < 5mm can be included if the investigator considers on clinical grounds that metastases are unlikely. Patients with multiple lung nodules should not be included unless there is a strong case that these do not represent metastases, e.g., stable on imaging for over 12 months, non-malignant aetiology apparent. The level of clinical suspicion may be influenced by clinical stage, e.g., N3 disease, low neck nodes. In general if there is any doubt patients should be excluded.
* Previous radical RT to the head & neck region, excluding superficial RT for a non-melanomatous skin cancer.
* Patients with prior cancers, except: those diagnosed > 5 years ago with no evidence of disease recurrence and clinical expectation of recurrence of less than 5%; or successfully treated non-melanoma skin cancer; or carcinoma in situ of the cervix.
* Significant intercurrent illness that will interfere with the chemotherapy or radiation therapy such as HIV infection, cardiac failure, pulmonary compromise, active infection
* Any history of myocardial infarction, ventricular arrhythmias, or unstable angina within the last 6 months
* Pregnant or lactating women.
* Weight loss greater than 20 % of usual body weight in the 3 months preceding trial entry
* High risk for poor compliance with therapy or follow up as assessed by the investigator
* Prior radiation to greater than 30% of the bone marrow
* Prior systemic chemotherapy for cancer
* Refusal by male or female patients, to use appropriate contraception during the study and for 3 months afterwards
* Any condition or circumstance which might prevent the patient being able to give valid informed consent, or from completing participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-04; Primary Completion 2014-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Safety and Feasibility | An initial 6 patients will be treated. Once all these patients have a 2 week post RT review there will be analysis. If <= 1 patient has a DLT than the treatment is deemed safe.

SECONDARY OUTCOMES:
Failure free survival (FFS) | All patients will be followed until the last patient enrolled has a minimum follow up of 2 years post treatment.
Time to local and/or regional failure | All patients will be followed until the last patient enrolled has a minimum follow up of 2 years post treatment.
Overall survival | All patients will be followed until the last patient enrolled has a minimum follow up of 2 years post treatment.
Site of first failure | All patients will be followed until the last patient enrolled has a minimum follow up of 2 years post treatment.
Acute and late treatment toxicities | All patients will be followed until the last patient enrolled has a minimum follow up of 2 years post treatment.

CONTACTS AND LOCATIONS:
Overall Officials: June Corry, Study Chair — Peter MacCallum Cancer Centre, Australia; Danny Rischin, Study Chair — Peter MacCallum Cancer Centre, Australia
Locations (1):
- Peter MacCallum Cancer Centre, Melbourne, Victoria, Australia

REFERENCES:
- See also: Click here for more information about this study on the TROG official website — http://www.trog.com.au